CLINICAL TRIAL: NCT01788657
Title: Internet-based Cognitive Behavior Therapy for Depression With Standard Treatment Material Compared to a Condensed Version
Brief Title: iCBT for Depression - Standard Versus Condensed Treatment Material
Acronym: KONRAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro County Council (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Fredrik Holländare, PhD, Örebro County Council
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dnr 63:2012
Record Dates: First submitted 2013-02-01; First posted 2013-02-11 (Estimated); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Major Depression
Keywords: Depression; Internet; Cognitive Behavior Therapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard internet-based cognitive behavior therapy (Experimental): Standard internet-based cognitive behavior therapy for depression with a written treatment material consisting of 60000 words (textmaterial only).
  Interventions: Behavioral: Standard internet-based cognitive behavior therapy
- Condensed internet-based cognitive behavior therapy (Experimental): Condensed internet-based cognitive behavior therapy for depression with a written treatment material consisting of 30000 words (available as text or audio).
  Interventions: Behavioral: Condensed internet-based cognitive behavior therapy

INTERVENTIONS:
Behavioral: Standard internet-based cognitive behavior therapy — Introduction to CBT and depression, Behavioral activation, Cognitive restructuring, Improve sleep, Handeling anxiety, Relapse prevention
  Other Names: Standard iCBT
  Arms: Standard internet-based cognitive behavior therapy
Behavioral: Condensed internet-based cognitive behavior therapy — Introduction to CBT and depression, Behavioral activation, Cognitive restructuring, Improve sleep, Handeling anxiety, Relapse prevention
  Other Names: Condensed iCBT
  Arms: Condensed internet-based cognitive behavior therapy

SUMMARY:
Internet-based cognitive behavior therapy (iCBT) has been shown effective for depression in several studies, however the investigators know very little about how the written treatment material should be designed to be effective and at the same time acceptable to the patients. The investigators are not aware of any research that has investigated if slow readers, or persons with difficulty concentrating, can use the standard material or if they would benefit more from using an adapted version.

In this study the investigators will assess reading speed and the ability to concentrate in all patients and then randomise them to an internet-based treatment for depression using either a standard material or a condensed one. The condensed material consists of 30000 words and will be available as text files and on audio files. The standard material consists of 60000 words and is only available as text files. Both groups will have the possibility of e-mail contact with a personal therapist during the treatment.

Patients will be recruited within Örebro County by referrals and self-referrals. The goal is to recruit between 200 and 300 patients during 2 years. The treatment time will be 10 weeks and all patients will be assessed for depression at an interview with a psychologist. There will also be interviews after treatment and one year after treatment. The most important outcome will be depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Fullfill criteria for diagnosis of major depression
* Being able to read and write Swedish
* Have access to the internet
* Being a resident in Örebro county

Exclusion Criteria:

* Severe depressive symptoms (>34 on the MADRS-S)
* High risk for suicide
* Attending cognitive behavior therapy
* Psychosis
* Bipolar disorder
* Addiction to alcohol or illegal drugs
* A somatic or psychiatric condition that is a contraindication for iCBT or in some way debars iCBT, or have to be treated before depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2013-10-29 (Actual); Primary Completion 2017-12-03 (Actual); Study Completion 2017-12-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms at post-treatment and after 12 months | At baseline, after 12 weeks, after 12 months
  Depressive symptoms will be measured by the self-report measure Montgomery-Åsberg Depression Rating Scale- self-rated.

SECONDARY OUTCOMES:
Change from baseline in diagnostic status for Major depression | Pre-treatment, after 12 weeks and after 1 year
  The diagnostic status (depression) will be assessed in a face-to-face interview using the structured material Mini-International Neuropsychiatric Interview (M.I.N.I.).
Change from baseline in symptoms of anxiety | Pre-treatment, after 12 weeks and after 1 year
  Symptoms of anxiety will be conducted using the self-report measure Beck Anxiety Inventory (BAI)
Post-treatment treatment satisfaction | After 12 weeks
  Post-treatment treatment satisfaction will be measured by the self-report measure Client Satisfaction Questionnaire (CSQ)
Therapist time | Post treatment
  Therapist time will be measured automatically by the IT-platform and assesses the time spent on each patient by each therapist. A mean time will be calculated to report an estimated time needed to treat one patient with the two interventions.
Alcohol use | Pre treatment
  To assess alkolhol use the AUDIT-questionnaire will be filled out at pre treatment.
Drug use | Pre treatment
  To assess drug use the DUDIT-questionnaire will be filled out at pre treatment.
Treatment satisfaction at follow up | After 1 year
  Treatment satisfaction at follow up will be measured by the self-report measure Client Satisfaction Questionnaire (CSQ)

OTHER OUTCOMES:
Reading speed | Pre treatment
  To assess reading speed the "Diagnostiskt Läs och Skrivprov" (DLS) will be administered during the pre treatment interview.
Ability to concentrate | Pre treatment
  To assess the ability to concentrate six items from the WHO adult scale for attention deficit disorder (ASRS-VI.I) will be administered during the pre treatment interview.
Change from baseline in risk for suicide | After 1,2,3,4,5,6,7,8,9,10,11,12 weeks
  Change in risk for suicide will be measured by item 9 in the MADRS-S every week

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Holländare, PhD, Principal Investigator — Örebro County Council
Locations (1):
- Örebro County Council, Örebro, Örebro County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Please contact us with suggestions for collaboration.
Supporting Information: Study Protocol, ICF, Analytic Code
Access Criteria: Upon request